CLINICAL TRIAL: NCT05903248
Title: Validity and Reliability of the Upper Extremity Star Balance Test in Amateur League American Football Players
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: American Football Players Star
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Athletic Injuries
Keywords: balance
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amateur American Football Team

SUMMARY:
American football is a team activity that calls for many difficult qualities, including speed, endurance, speed, strength, and quickness. It is getting more and more popular among professional and amateur players, particularly in our nation.

DETAILED DESCRIPTION:
Balance is defined as maintaining posture and postural continuity throughout a movement, despite a changing environment or condition while the body is in motion.

However, the upper extremity star balancing test offers information on only three access elements and the possible dangers may not be thoroughly assessed. As a more thorough upper extremity dynamic balance test, the upper extremity star balance test can provide data in eight directions of physicians and physiotherapists and coaches.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals between the ages of 18-25
* Being an American football player
* Regular attendance at training sessions

Exclusion Criteria:

* Known neurological disorder
* Serious orthopedic disorders that prevent exercise
* cognitive impairment

Ages: 18 Years to 25 Years | Sex: Male
Age Groups: Adult
Study Population: Bahcehir University Amateur Football Team players will participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-21 (Estimated); Primary Completion 2023-06-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Star Excursion Balance Test | one day
  Eight directions including anterior, superomedial, medial, inferomedial, posterior, inferolateral, lateral, and superolateral were marked on floor by tapes with scale and the angle between each strip of tape were 45°. The minimum unit of the UESEBT was 0.5 cm. Distances for analysis were normalized by dividing the right upper limb length of every participant, and then multiplying by 100.
Sitting Medicine Ball Throwing | one day
  Throwing Medicine Ball: Individuals will be asked to take a position in front of a wall, with their feet shoulder-width apart, to grasp the medicine ball with both hands. A medicine ball weighing two kg will be used in this test. Individuals will be asked to bring the medicine ball to the head level and throw it forward. The thrown distance is recorded.
Push Up Test. | one day
  The push-up test was performed with the participant pushing their arms off the floor until their elbows were straight while keeping their legs and back straight. This movement was repeated as many times as possible, ending when the subject stopped or the participant did not perform the push-ups properly or held the correct position several times.
Closed Kinetic Chain Upper Extremity Stability Test (TEST) | one day
  Individuals were positioned in the push-up position, with their bodies aligned in a straight line when viewed from the side, with a distance of 90 cm between their hands. The athletes were asked to touch the dorsum of the dominant hand and the other hand within 15 seconds, and the total number of repetitions was recorded.
Upper extremity Y Test | one day
  Upper extremity lengths are determined by measuring the distance between the C7 cervical vertebra processus spinosus and the middle fingertip of the athletes. In this position, the athletes are positioned perpendicular to the middle extension of the Y balance kit (the arm that makes an angle of 135° with the other ends). Afterwards, the athlete is asked to push the platform apparatus along the superior and inferior arms, which are lateral to the lateral side of his fixed hand, and take it to the last point it can take. Y balance scores were found using the reach distance and limb length in each direction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu HR, Zhang YH, Mao Y, Ngo TL, Zhang Q, He G, Feng Z, Sun W, Wang XQ. Validity and reliability of upper extremity star excursion balance test in adolescent swimmers. J Exerc Sci Fit. 2023 Apr;21(2):210-217. doi: 10.1016/j.jesf.2023.02.003. Epub 2023 Feb 27. PMID 36923209